CLINICAL TRIAL: NCT03768752
Title: Left Ventricular Diastolic Dysfunction as a Risk Factor for Interstitial Lung Edema in Septic Patients on the Intensive Care Unit
Brief Title: Diastolic Dysfunction and Interstitial Lung Edema in Septic Patients
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Ursula Kahl, Dr. med., Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: DD-Sepsis
Record Dates: First submitted 2018-11-30; First posted 2018-12-07 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Sepsis; Diastolic Dysfunction; Lung Edema; Fluid Overload
Keywords: intensive care unit; echocardiography
MeSH Terms: conditions — Sepsis; Pulmonary Edema; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diastolic Dysfunction: Patients with pre-existing or new diastolic dysfunction.
- Normal Diastolic Function: Patients with normal diastolic function.

SUMMARY:
Sepsis is one of the most challenging conditions with an exceptionally high mortality rate. Diastolic Dysfunction is common in septic patients and has been found to be associated with mortality. However, the reasons for this remain unclear. Therefore, the goal of this study is to investigate diastolic dysfunction in septic patients on the intensive care unit. Special attention is paid to the presence of lung edema and general edema as a potential link between diastolic dysfunction and elevated mortality in septic patients. During the septic phase daily ultrasound examinations of heart and lung will be performed as to monitor diastolic function and lung edema.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the intensive care unit diagnosed with SIRS (systemic inflammatory response syndrome) or Sepsis.

Exclusion Criteria:

* Patients with hemodynamically relevant cardiac defects.
* Patients with mitral valve replacement.
* Patients with pericardial effusion.
* Patients with atrial fibrillation.
* Patients with pacemaker therapy.
* Patients with BMI > 35 kg/m2.
* Patients with poor examination conditions for ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on the intensive care unit of the university hospital Hamburg-Eppendorf diagnosed with sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Diastolic Dysfunction | While in septic condition, up to 10 days maximum.
  Diastolic Dysfunction specified by echocardiographic doppler derived mitral inflow pattern and tissue doppler derived diastolic mitral annular velocities (E/E').
Pulmonary Edema | While in septic condition, up to 10 days maximum.
  Pulmonary edema specified by B line ultrasound score (Lung ultrasound protocol for the assessment of pulmonary fluid status according to Enghardt et al. 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Kahl, MD, Principal Investigator — Klinik und Poliklinik für Anästhesie Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätskrankenhaus Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleischmann C, Scherag A, Adhikari NK, Hartog CS, Tsaganos T, Schlattmann P, Angus DC, Reinhart K; International Forum of Acute Care Trialists. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016 Feb 1;193(3):259-72. doi: 10.1164/rccm.201504-0781OC. PMID 26414292
- [Background] Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med. 2003 Apr 17;348(16):1546-54. doi: 10.1056/NEJMoa022139. PMID 12700374
- [Background] Sanfilippo F, Corredor C, Fletcher N, Landesberg G, Benedetto U, Foex P, Cecconi M. Diastolic dysfunction and mortality in septic patients: a systematic review and meta-analysis. Intensive Care Med. 2015 Jun;41(6):1004-13. doi: 10.1007/s00134-015-3748-7. Epub 2015 Mar 24. PMID 25800584
- [Background] Enghard P, Rademacher S, Nee J, Hasper D, Engert U, Jorres A, Kruse JM. Simplified lung ultrasound protocol shows excellent prediction of extravascular lung water in ventilated intensive care patients. Crit Care. 2015 Feb 6;19(1):36. doi: 10.1186/s13054-015-0756-5. PMID 25656060
- [Background] Suehiro K, Morikage N, Murakami M, Yamashita O, Samura M, Hamano K. Significance of ultrasound examination of skin and subcutaneous tissue in secondary lower extremity lymphedema. Ann Vasc Dis. 2013;6(2):180-8. doi: 10.3400/avd.oa.12.00102. Epub 2013 May 10. PMID 23825499
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Derived] Kahl U, Schirren L, Yu Y, Lezius S, Fischer M, Menke M, Sinning C, Nierhaus A, Vens M, Zollner C, Kluge S, Goepfert MS, Roeher K. Left Ventricular Diastolic Dysfunction Is Not Associated With Pulmonary Edema in Septic Patients. A Prospective Observational Cohort Study. Front Cardiovasc Med. 2022 Jul 1;9:900850. doi: 10.3389/fcvm.2022.900850. eCollection 2022. PMID 35845063